CLINICAL TRIAL: NCT05416710
Title: Prospective Community Cancer Clinics-based Approach to Optimize Germline Testing in Cancer Patients in Rural Setting to Address Racial Disparities: UNIversal Germline Testing in the communitY (UNITY) Study
Brief Title: Universal Germline Testing in the Community
Acronym: UNITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Invitae Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-001-017
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Cancer; Solid Tumor; Solid Tumor, Adult
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained as baseline for germline genetic testing (1 EDTA Tube with 4-7mL of blood) and future research use (2 Streck tubes for 20mL of blood total).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Solid tumor cancers: Adult participants with a diagnosis of a solid tumor cancer who are able to consent to the study and who are interested in undergoing germline genetic testing will receive testing using Invitae's 84 gene Multi-Cancer panel.
  Interventions: Diagnostic Test: Invitae's 84 gene multi-cancer panel.

INTERVENTIONS:
Diagnostic Test: Invitae's 84 gene multi-cancer panel. — Invitae's Multi-Cancer panel analyzes 84 genes associated with hereditary cancers across major organ systems.

SUMMARY:
This study seeks to enroll participants who have a diagnosis of a solid tumor cancer and are willing to undergo germline genetic testing for cancer risk. At baseline, patients will be asked to provide 2 types of blood samples: 1 tube for clinical genetic testing and 2 tubes for future research use. A tumor sample from a previous resection or biopsy will also be obtained and sent to the sponsor. The clinician will be asked to provide relevant medical history and demographic information to the sponsor in the form of electronic case report forms.

DETAILED DESCRIPTION:
This study seeks to enroll adult participants who have a diagnosis of a solid tumor cancer and are willing to undergo germline genetic testing for cancer risk using Invitae's Multi-Cancer gene panel. At baseline, patients will be asked to provide 2 types of blood samples: 1 tube for clinical genetic testing and 2 tubes for future research use. A tumor sample from a previous resection or biopsy will also be obtained and sent to the sponsor. The participant's clinician will be asked to provide relevant medical history and demographic information to the sponsor in the form of electronic case report forms at 3 timepoints: 1 month following the results of the participants genetic testing, one year post genetic testing, and 2 years post genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient has consented to germline genetic testing
* Patient has a histologically confirmed diagnosis of a solid tumor cancer
* Patient is willing to release previously collected tissue sample
* Patient is willing to provide research blood samples
* Patient must be at least 18 years of age

Exclusion Criteria:

* Patient is unable to consent.
* Patient with hematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with solid tumor cancer who are willing to undergo germline genetic testing and who can consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Pathogenic Germline Variants (PGV) | Will be assessed at baseline only.
  Assess rate of PGVs in the trial participants using Invitae's 84 gene multi-cancer gene panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Blood and Cancer Care Associates, PA', Rock Hill, South Carolina, United States